CLINICAL TRIAL: NCT04286997
Title: VARA: Motor Rehabilitation Protocol With GRAIL for Patients Affected by Hemiparesis
Brief Title: VARA (Virtual and Augmented Reality Applications in Rehabilitation): Motor Rehabilitation Protocol With GRAIL for Patients Affected by Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 585
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Hemiparesis
Keywords: GRAIL; children; rehabilitation; virtual reality; hemiparesis
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GRAIL population (Experimental): patients are treated with 20 sessions of GRAIL rehabilitation, associated to 20 traditional physiotherapy sessions (1+1 a day, during a period of 30 days)
  Interventions: Device: GRAIL population
- traditional population (Active Comparator): subjects are treated with 40 sessions of traditional physiotherapy (2 a day, during a period of 30 days)
  Interventions: Device: GRAIL population

INTERVENTIONS:
Device: GRAIL population — each subjects included in the intervention group will receive 20 GRAIL sessions, aimed to the walking pattern improvement, associated with 20 traditional physiotherapy sessions, aimed to the stabilization of the trained competences

SUMMARY:
The main goal of the study is to verify the efficacy of the GRAIL system in respect to the walking pattern improvement in a population of hemiparetic subjects.

In particular, the specific goals will be:

* increase in walking symmetry and a better distribution among the time of stance and swing.
* Kinematics and Kinetics correction, with incentive of more corrected activation timing.
* Recruitment of the muscles most involved by the paresis, with the help of visual feedback.
* walking speed increase (but with the priority of the walking pattern)
* increase in the resistance
* Stregthening of the support reaction

ELIGIBILITY:
Inclusion Criteria:

* hemiparetic patients as a consequence of acquired brain injury

Exclusion Criteria:

* excessive muscular spasticity or contractures.
* recent (under 6 months) lower limbs surgery
* cognitive or emotional/relational obstacles to the therapy

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Gait Analysis | 1 month
  Analysis of the walking pattern performed with traditional gait analysis lab and with GRAIL system
Gross Motor Functional Movement | 1 month
  Assessment of the kinetic function, divided into 5 dimensions, range from 0 to 88, 0 meaning worse scores and 88 healthy subjects.

SECONDARY OUTCOMES:
6 Minute Walking Test | 1 month
  recording of the distance run by the patient in a lapse of time of 6 minutes
Functional Assessment Questionaire | 1 month
  Questionaire Filled in by the patients or by the parents, on the perception of the walking ability, range from 1 (subjects unable to step) to 10 (healthy subjects)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS E.Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No